CLINICAL TRIAL: NCT07042581
Title: Evaluation of Revaree Plus in Women With Breast Cancer
Brief Title: A Study of Revaree Plus in People With Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-374
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Stage 0 Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; Stage 0 Breast Carcinoma; Stage II Breast Carcinoma; Stage III Breast Carcinoma; Hormone-receptor-positive Breast Cancer; Hormone Receptor Positive Breast Carcinoma; Hormone Receptor Positive Malignant Neoplasm of Breast
Keywords: Breast Cancer; Stage 0 Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; Stage 0 hormone receptor positive breast cancer; Stage I hormone receptor positive breast cancer; Stage II hormone receptor positive breast cancer; Stage III hormone receptor positive breast cancer; Revaree; 24-374; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hormone-receptor positive breast cancer participants (Experimental): Participants will have a diagnosis of Stage 0-III Hormone-receptor positive breast cancer
  Interventions: Drug: Revaree Plus

INTERVENTIONS:
Drug: Revaree Plus — Revaree Plus is a hyaluronic acid vaginal suppository

SUMMARY:
The purpose of this study is to find out whether Revaree Plus is effective at improving vaginal health for people who are having symptoms of vaginal dryness during breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing informed consent.
* Stage 0-3 hormone-receptor positive breast cancer confirmed at MSKCC
* Able to complete study questionnaires in English or Spanish
* Breast cancer patients must have completed primary therapy (surgery, and/or chemotherapy, and/or radiation therapy) or currently on maintenance therapy
* Currently on an aromatase inhibitor or tamoxifen or Selective Estrogen Receptor Modulators (SERM)
* Currently have no clinical evidence of disease
* Reporting being bothered by vaginal symptoms of estrogen deprivation (i.e., vaginal dryness, dyspareunia, or discomfort [pain with intercourse or examination])
* A total score of 4 or greater in VAS
* Without history of other cancers (excluding non-melanoma skin cancer)
* Must sign an informed consent indicating that the participant understands the purpose of, and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* Inability to provide informed consent
* Vaginal bleeding of unknown etiology within 12 months of study entry
* Currently taking hormone replacement therapy [local or systemic] (Patients must discontinue for 4 weeks in order to be eligible prior to study enrollment)
* Existing use of external estrogens or nonhormonal moisturizers (Patients must discontinue for 4 weeks in order to be eligible prior to study enrollment)
* No known allergies to any ingredients in 10mg HLA suppository

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2029-06-20 (Estimated); Study Completion 2029-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Vaginal Assessment Scale from baseline to 8 weeks | 8 weeks
  The primary study objective is to evaluate whether vaginal health improves from baseline to 8 weeks of treatment with Revaree Plus as measured by the Vaginal Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk-Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org